CLINICAL TRIAL: NCT06152757
Title: Clinical Study on the Safety and Preliminary Efficacy of BGT007H Cell Therapy in Patients With Recurrent/Refractory Gastrointestinal Tumors
Brief Title: BGT007H Cells for the Treatment of Recurrent/Refractory Gastrointestinal Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR-BGT-003
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Tumors
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGT007H injection (Experimental): Intravenous infusion
  Interventions: Biological: First dose; Biological: Second dose; Biological: The third dose; Biological: The fourth dose

INTERVENTIONS:
Biological: First dose — 1.0×10^8cells,Intravenous infusion，1 subject is planned to be enrolled
Biological: Second dose — 3.0×10^8cells,Intravenous infusion，3 subject is planned to be enrolled
Biological: The third dose — 1.0×10^9cells,Intravenous infusion，3 subject is planned to be enrolled
Biological: The fourth dose — 3.0×10^9cells,Intravenous infusion，3 subject is planned to be enrolled

SUMMARY:
This study is an exploratory single-arm, open, modified "3+3" dose escalation study with BGT007H injection. Approximately 11 to 14 subjects with recurrent/refractory gastrointestinal tumors will be enrolled to evaluate the safety of BGT007H injection.

Four dose levels were designed for this study: 1.0×10^8cells, 3.0×10^8cells, 1.0×10^9cells, and 3.0×10^9cells. The primary objective of this study was to evaluate the safety, tolerability and pharmacokinetic profile of BGT007H cell therapy in patients with recurrent/refractory digestive tract tumors, to determine the maximum tolerated dose or the best effective dose, and to initially evaluate the effectiveness of BGT007H cell products.

DETAILED DESCRIPTION:
Main research objectives:

Evaluation of the safety and tolerability of BGT007H cell therapy in patients with recurrent/refractory gastrointestinal tumors

Secondary research objectives:

1. Evaluate the pharmacokinetic (PK) characteristics of BGT007H cells after reinfusion;
2. Evaluation of the initial effectiveness of BGT007H cell therapy in patients with recurrent/refractory gastrointestinal tumors

Exploratory Purpose

1. Exploring the correlation between the proliferation and survival of BGT007H cells in vivo and their therapeutic effects;
2. Exploring the correlation between target expression levels and efficacy

ELIGIBILITY:
Inclusion Criteria:

* 1. Resources sign written informed consent;
* 2, age ≥18, male and female can;
* 3. Expected survival ≥3 months;
* 4. The Eastern Cancer Collaboration (ECOG) physical status score was 0-1;
* 5. Biopsy specimen or pathological wax section test (within 3 years before accepting the signed informed consent) : positive target test;
* 6. According to RECISTv1.1 solid tumor evaluation criteria, there is at least one measurable lesion;
* 7. Patients with advanced gastrointestinal tumors (esophageal cancer, gastric cancer, pancreatic cancer or colorectal cancer, etc.) who have been diagnosed by histology/cytology as having failed the standard of second-line or above treatment or are not suitable for/refuse to accept the standard treatment or cannot tolerate the standard treatment; The definition of intolerance: according to CTCAE V5.0, the occurrence of ≥Ⅳ hematological toxicity or ≥Ⅲ non-hematological toxicity or ≥Ⅱ damage to the heart, liver, kidney and other important organs during treatment; Treatment failure is defined as disease progression (PD) during treatment or recurrence after the end of treatment (including postoperative recurrence);
* 8, can establish monopexy or venous blood collection venous access, and there are no other contraindications for blood cell separation;
* 9, with adequate organ and bone marrow function;
* 10. During the study period and for 6 months after the end of dosing, fertile subjects (both male and female) must use effective medical contraception. For female subjects of reproductive age, a pregnancy test should be performed within 72 hours before the first dose, and the result is negative.

Exclusion Criteria:

* 1. Active central nervous system metastasis (except stable after treatment);
* 2, HIV positive, HBsAg positive simultaneously detected HBV DNA copy number positive (quantitative detection ≥1000cps/ml), HCV antibody positive and HCV RNA positive;
* 3, mental or mental illness can not cooperate with treatment and efficacy evaluation;
* 4. Subjects with severe autoimmune diseases and long-term use of immunosuppressants;
* 5. Active or uncontrollable infection requiring systemic treatment within 14 days prior to enrollment;
* 6. Any unstable systemic disease (including but not limited to: Active infections (except local infections); Unstable angina pectoris Cerebral ischemia or cerebrovascular accident (within 6 months prior to screening) Myocardial infarction (within 6 months prior to screening) Congestive heart failure (New York Heart Association [NYHA] classification ≥Ⅲ; Severe arrhythmias requiring medical treatment; Have heart disease that requires treatment or uncontrolled hypertension after treatment (blood pressure > 160mmHg/100mmHg);
* 7, combined with lung, brain, kidney and other important organ dysfunction;
* 8. The subject has undergone major surgery or severe trauma within 4 weeks prior to receiving cell therapy, or is expected to undergo major surgery during the study period;
* 9. Received any systemic chemotherapy, immunotherapy or small molecule targeted therapy within 1-2 weeks or 5 half-lives (whichever is shorter) before anapheresis;
* 10. The subject currently has or has had other malignant tumors that cannot be cured within 3 years, except cervical cancer or basal cell carcinoma of the skin, and other malignant tumors with a disease-free survival of more than 5 years;
* 11, received chimeric antigen receptor modified T cells (including CAR-T, CTT-T) treatment within half a year;
* 12. Combined graft-versus-host disease (GVHD)
* 13. Subjects who were receiving systemic steroid therapy prior to screening and who were determined by the investigator to require long-term use of systemic steroid therapy during treatment (except for inhalation or topical use); And subjects treated with systemic steroids within 72 hours prior to cell transfusion (except for inhalation or topical use);
* 14. Severe allergy or history of allergy;
* 15. Subjects requiring anticoagulation therapy;
* 16, pregnant or breastfeeding women, or six months within the pregnancy plan (unisex;
* 17. Researchers believe that there are other reasons for not being included in the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-07-19 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | From the infusion (Day 0) to Day 28
  Incidence of adverse events defined as Dose-Limiting Toxicity (DLT).
Maximum tolerated dose | From the infusion (Day 0) to Day 28
  The maximum CAR-T dose that can be tolerated in the study.
AE, SAE, AESI, CRS, ICANS, TEAE | The day of leukapheresis to 12 months after infusion
  The incidence of adverse events (AE), serious adverse events (SAE), adverse events of special interest (AESI), cytokine release syndrome (CRS) immune cell associated neurotoxicity syndrome (ICANS) and treatment-emergent adverse events (TEAE).

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China